CLINICAL TRIAL: NCT05447078
Title: Impact of Oral Immulina TM on Natural Killer Cell Activities and Other Biomarkers Associated With Increasing Host Immune Resilience to Upper Respiratory Viruses in Normal Human Volunteers
Brief Title: Spirulina Oral Supplement for Enhancing Host Resilience to Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2020-0020; 1U19AT010838-01 (NIH)
Record Dates: First submitted 2022-06-21; First posted 2022-07-07 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Immulina TM; Natural Killer Cells (NK); Botanical Dietary Supplement; Influenza; Dietary Supplementation
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): inert capsules; 2 capsules given by mouth in the morning and 2 capsules given by mouth in the evening for 16 weeks duration.
  Interventions: Dietary Supplement: Placebo
- Immulina TM 200 mg/day (Experimental): Immulina Dietary supplementation (200 mg per capsule); 1-200 mg capsule and 1 placebo capsule given by mouth in the morning and 2 placebo capsules given by mouth in the evening for 16 weeks duration.
  Interventions: Drug: Immulina TM
- Immulina TM 400 mg/day (Experimental): Immulina Dietary supplementation (200 mg per capsule); 1-200 mg capsule and 1 placebo capsule given by mouth in the morning and 1-200 mg capsule and 1 placebo capsule given by mouth in the evening for 16 weeks duration.
  Interventions: Drug: Immulina TM
- Immulina TM 800 mg/day (Experimental): Immulina Dietary supplementation (200 mg per capsule); 2-200 mg capsules given by mouth in the morning and 2-200 mg capsules given by mouth in the evening for 16 weeks duration.
  Interventions: Drug: Immulina TM

INTERVENTIONS:
Drug: Immulina TM — Immulina TM is a highly standardized extract derived from various preparations of Spirulina, a cyanobacterium, marketed as a dietary supplement and has been utilized in several clinical studies describing its immunopotentiating properties.
  Other Names: Spirulina
  Arms: Immulina TM 200 mg/day; Immulina TM 400 mg/day; Immulina TM 800 mg/day
Dietary Supplement: Placebo — Placebo is inert powder in cellulose capsule that appears identical to Immulina TM capsules.
  Arms: Placebo

SUMMARY:
This randomized, double blind, placebo controlled study aims to establish the impact of the oral supplement, Immulina TM, on enhancing host resilience to the effects of viral influenza infection in humans.

DETAILED DESCRIPTION:
This randomized, double blind, placebo controlled study aims to establish the impact of the oral supplement, Immulina TM, on increasing host resilience against the pathogenic effects of influenza virus infection in normal and immune compromised individuals by measuring a biomarker profile designed to reflect immune components associated with antiviral natural killer cell numbers and activity, cytotoxic T cell numbers, vaccine-related flu-specific antibody responses and cytokine profiles associated with host antiviral innate and adaptive immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-59 (study group 1) or ages 65 and above (study group 2)
* Any chronic illness must be determined (by PI team) to be stable as evidenced by no changes in medical regimens within 30 days of enrollment.
* Ability to comprehend the specific activities required to participate in the trial for which the participant is to be enrolled.

Exclusion Criteria:

* Any acute illness or significant injury within 30 days of enrollment.
* Specific disease entities, which, in the opinion of the PI, could reasonably be assumed to have dysfunctional immune function as a component of their illness. These include HIV, AIDS, uncontrolled asthma, uncontrolled eczema, uncontrolled allergic rhinitis, uncontrolled urticaria, Rheumatoid arthritis, lupus, inflammatory bowel disease, multiple sclerosis, Type-1 diabetes mellitus, Guillain-Barr syndrome, Grave's disease, Hashimoto's thyroiditis, myasthenia gravis or vasculitis.
* Active autoimmune diseases regardless of clinical stability. A history of autoimmune disease that is not considered active (i.e. no medical therapy for at least 1 year prior to enrollment) will not be excluded.
* History of unstable chronic illness within 30 days of enrollment.
* Unable/unwilling to commit to multiple research clinic visits which will be described in detail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Natural Killer cell (NK)-mediated cytotoxicity | 20 weeks
  NK cell-mediated cytotoxicity is characterized by cytolysis of a CFSE-labeled target cell (K562) by effector cells (NK cells). Labeled K562 are cultured with NK cells for a period of time, then all cells labeled with a live-dead stain, 7-AAD. The cytolytic activity is expressed as the percent dead K562.
  Differences in cytolytic activity (% dead K562) from baseline to 20 weeks.

SECONDARY OUTCOMES:
Natural Killer (NK) cell count | 20 weeks
  Differences in NK cell counts from baseline to 20 weeks
Cytotoxic T lymphocyte (CTL) number | 20 weeks
  Differences in CTL counts from baseline to 20 weeks
Plasma cytokine profile; IL1b, IL6, TNF alpha, IL2, IL7, IL12, IL15 and IL18; pg/mL | 20 weeks
  Differences in plasma cytokine profiles from baseline to 20 weeks
Immunophenotyping panel biomarkers- CD3, CD4, CD8, CD25, FoxP3, IL10, Interferon gamma, IL4, TGF beta counts | 20 weeks
  CD3 (mature T cells), CD4(T helper/inducer cell), CD8 (T suppressor/cytotoxic cell), CD25 (IL2 suppressor), FoxP3 (T regulator cell), IL10 (T regulatory suppressor cell), Interferon gamma (T helper 1 cell), IL4 (T helper 2 cell) and TGF beta (T regulatory suppressor cell) counts in human peripheral blood mononuclear cells measured by flow cytometry.
  Differences in Immunophenotyping panel biomarker counts from baseline to 20 weeks
Influenza A IgG antibody, U/mL | 20 weeks
  Differences in Influenza A IgG antibody U/mL from baseline to 20 weeks
Influenza B IgG antibody, U/mL | 20 weeks
  Differences in Influenza B IgG antibody U/mL from baseline to 20 weeks
serum Interferon gamma, pg/mL | 20 weeks
  Differences in Interferon gamma levels from baseline to 20 weeks
serum Interferon alpha, pg/mL | 20 weeks
  Differences in Interferon alpha levels from baseline to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D Marshall Jr., MD, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No